CLINICAL TRIAL: NCT04915950
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Assess the Effect of Oral Temanogrel on Digital Blood Flow in Subjects With Raynaud's Phenomenon Secondary to Systemic Sclerosis
Brief Title: A Study to Assess the Effect of Oral Temanogrel on Digital Blood Flow in Adult Participants With Raynaud's Phenomenon Secondary to Systemic Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: APD791-204; C5071001 (Other: Alias Study Number)
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Raynaud's Phenomenon Secondary to Systemic Sclerosis
Keywords: Raynaud's phenomenon; SSc-RP; Systemic sclerosis; SSc; Digital cold sensitivity; Digital blood flow; APD791; Temanogrel
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic | interventions — APD791

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Temanogrel (Stage A Dose 1) (Experimental)
  Interventions: Drug: Temanogrel
- Temanogrel (Stage A Dose 2) (Experimental)
  Interventions: Drug: Temanogrel
- Placebo (Stage A) (Placebo Comparator)
  Interventions: Drug: Placebo
- Temanogrel (Stage B Dose 1) (Experimental)
  Interventions: Drug: Temanogrel
- Temanogrel (Stage B Dose 2) (Experimental)
  Interventions: Drug: Temanogrel
- Placebo (Stage B) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Temanogrel — Participants will receive a single oral dose of temanogrel during the treatment visit.
  Other Names: APD791
  Arms: Temanogrel (Stage A Dose 1); Temanogrel (Stage A Dose 2); Temanogrel (Stage B Dose 1); Temanogrel (Stage B Dose 2)
Drug: Placebo — Participants will receive a single oral dose of temanogrel matching placebo during the treatment visit.
  Arms: Placebo (Stage A); Placebo (Stage B)

SUMMARY:
The purpose of this study is to determine whether oral temanogrel improves digital blood flow in participants with Raynaud's phenomenon secondary to systemic sclerosis (SSc-RP) as a potential safe and effective treatment for symptoms associated with SSc-RP.

DETAILED DESCRIPTION:
The study will be conducted in 2 stages: Stage A and Stage B. In both stages, participants will be equally randomized in a double-blind manner to a 3-period crossover treatment sequence. Separate cohorts of participants will participate in each stage. In Stage A, participants will be treated with two dose levels of temanogrel and placebo. Doses in Stage B will be determined based on the results of Stage A.

ELIGIBILITY:
Inclusion Criteria:

* Raynaud's phenomenon (defined as a history of digital cold sensitivity associated with color changes of cyanosis and pallor, with on average at least 5 attacks per week during the winter period) secondary to systemic sclerosis (SSc)
* Both men and women participants agree to use a highly effective method of birth control if the possibility of conception exists
* Body mass index 18.0 to 40.0 kilograms per square meter (kg/m^2), inclusive

Exclusion Criteria:

* Active digital ulcer(s), recent history (within 3 months of Screening) of digital ulcers, or history of recurrent digital ulcerations that in the opinion of the Investigator increase the likelihood of developing a digital ulcer during the course of the study. Any history of gangrene, amputations, or other critical digital ischemic event
* Raynaud's phenomenon due to any cause other than SSc
* Severe gastrointestinal complications related to SSc that in the opinion of the Investigator could significantly affect study drug absorption
* History of gastrointestinal bleeding or active gastric or duodenal ulcers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - UPMC Arthritis and Auotimmune Clinic, Pittsburgh, Pennsylvania
- United Kingdom (3):
  - Ninewells Hospital & Medical School, Dundee, Scotland
  - Royal United Hospitals Bath, Bath
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD791-204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned to be conducted in 2 stages: Stage A and Stage B. Stage B was not conducted due to early termination of the study.
Pre-assignment Details: A total of 13 participants were enrolled and randomized in the study.
Groups:
- Temanogrel 120 mg Then Temanogrel 60 mg Then Placebo: Participants received oral temanogrel 120 milligram (mg) (6 temanogrel capsules of 20 mg) once per treatment visit (A) orally once on Day 1 of treatment period 1. Period 1 was followed by treatment period 2. On Day 1 of treatment period 2, participants received temanogrel 60mg (3 temanogrel capsules of 20 mg each and 3 capsules of placebo) once orally (B). Period 2 was followed by treatment period 3. On Day 1 of treatment period 3, participants received placebo matched to temanogrel capsules (6 capsules) once orally (C). Study treatment administrations between two periods were separated by washout period of at least 72 hours to 7 days.
- Temanogrel 120 mg Then Placebo Then Temanogrel 60mg: Participants received oral temanogrel 120 mg (6 temanogrel capsules of 20 mg) once per treatment visit (A) orally once on Day 1 of treatment period 1. Period 1 was followed by treatment period 2. On Day 1 of treatment period 2, participants received placebo matched to temanogrel capsules (6 capsules) once orally (C). Period 2 was followed by treatment period 3. On Day 1 of treatment period 3, participants received participants received temanogrel 60mg (3 temanogrel capsules of 20 mg each and 3 capsules of placebo) once orally (B). Study treatment administrations between two periods were separated by washout period of at least 72 hours to 7 days.
- Temanogrel 60 mg Then Temanogrel 120 mg Then Placebo: Participants received temanogrel 60 mg (3 temanogrel capsules of 20 mg each and 3 capsules of placebo) once orally during treatment period 1 (B). Period 1 was followed by treatment period 2. On Day 1 of treatment period 2, participants received oral temanogrel 120 mg (6 temanogrel capsules of 20 mg) once per treatment visit (A) orally once on Day 1 of period 2. Period 2 was followed by treatment period 3. On Day 1 of treatment period 3, participants received placebo matched to temanogrel capsules (6 capsules) once orally (C). Study treatment administrations between two periods were separated by washout period of at least 72 hours to 7 days.
- Temanogrel 60 mg Then Placebo Then Temanogrel 120 mg: Participants received temanogrel 60mg (3 temanogrel capsules of 20 mg each and 3 capsules of placebo) once orally during treatment period 1 (B). Period 1 was followed by treatment period 2. On Day 1 of treatment period 2, participants received placebo matched to temanogrel capsules (6 capsules) once orally (C). Period 2 was followed by treatment period 3. On Day 1 of treatment period 3, participants received oral temanogrel 120 mg (6 temanogrel capsules of 20 mg) once per treatment visit (A) orally once on Day 1 of treatment period 3. Study treatment administrations between two periods were separated by washout period of at least 72 hours to 7 days.
- Placebo Then Temanogrel 120 mg Then Temanogrel 60 mg: Participants received placebo matched to temanogrel capsules (6 capsules) once orally (C). Period 1 was followed by treatment period 2. On Day 1 of treatment period 2, participants received oral temanogrel 120 mg (6 temanogrel capsules of 20 mg) once per treatment visit (A) orally once on Day 1 of period 2. Period 2 was followed by treatment period 3. On Day 1 of treatment period 3, participants received temanogrel 60 mg (3 temanogrel capsules of 20 mg each and 3 capsules of placebo) once orally (B). Study treatment administrations between two periods were separated by washout period of at least 72 hours to 7 days.
- Placebo Then Temanogrel 60 mg Then Temanogrel 120 mg: Participants received placebo matched to temanogrel capsules (6 capsules) once orally (C). Period 1 was followed by treatment period 2. On Day 1 of treatment period 2, participants received temanogrel 60mg (3 temanogrel capsules of 20 mg each and 3 capsules of placebo) once orally (B). Period 2 was followed by treatment period 3. On Day 1 of treatment period 3, participants received oral temanogrel 120 mg (6 temanogrel capsules of 20 mg) once per treatment visit (A) orally once on Day 1 of treatment period 3. Study treatment administrations between two periods were separated by washout period of at least 72 hours to 7 days.
Period: Stage A: Treatment Period 1 (1 Day)
Arm/Group | Temanogrel 120 mg Then Temanogrel 60 mg Then Placebo | Temanogrel 120 mg Then Placebo Then Temanogrel 60mg | Temanogrel 60 mg Then Temanogrel 120 mg Then Placebo | Temanogrel 60 mg Then Placebo Then Temanogrel 120 mg | Placebo Then Temanogrel 120 mg Then Temanogrel 60 mg | Placebo Then Temanogrel 60 mg Then Temanogrel 120 mg
Started | 2 | 2 | 2 | 2 | 3 | 2
Completed | 2 | 2 | 2 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage A:Washout Period(72hours to 7days)
Arm/Group | Temanogrel 120 mg Then Temanogrel 60 mg Then Placebo | Temanogrel 120 mg Then Placebo Then Temanogrel 60mg | Temanogrel 60 mg Then Temanogrel 120 mg Then Placebo | Temanogrel 60 mg Then Placebo Then Temanogrel 120 mg | Placebo Then Temanogrel 120 mg Then Temanogrel 60 mg | Placebo Then Temanogrel 60 mg Then Temanogrel 120 mg
Started | 2 | 2 | 2 | 2 | 3 | 2
Completed | 2 | 2 | 2 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage A: Treatment Period 2 (1 Day)
Arm/Group | Temanogrel 120 mg Then Temanogrel 60 mg Then Placebo | Temanogrel 120 mg Then Placebo Then Temanogrel 60mg | Temanogrel 60 mg Then Temanogrel 120 mg Then Placebo | Temanogrel 60 mg Then Placebo Then Temanogrel 120 mg | Placebo Then Temanogrel 120 mg Then Temanogrel 60 mg | Placebo Then Temanogrel 60 mg Then Temanogrel 120 mg
Started | 2 | 2 | 2 | 2 | 3 | 2
Completed | 2 | 2 | 2 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage A:Washout Period(72hours to 7days)
Arm/Group | Temanogrel 120 mg Then Temanogrel 60 mg Then Placebo | Temanogrel 120 mg Then Placebo Then Temanogrel 60mg | Temanogrel 60 mg Then Temanogrel 120 mg Then Placebo | Temanogrel 60 mg Then Placebo Then Temanogrel 120 mg | Placebo Then Temanogrel 120 mg Then Temanogrel 60 mg | Placebo Then Temanogrel 60 mg Then Temanogrel 120 mg
Started | 2 | 2 | 2 | 2 | 3 | 2
Completed | 2 | 2 | 2 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage A: Treatment Period 3 (1 Day)
Arm/Group | Temanogrel 120 mg Then Temanogrel 60 mg Then Placebo | Temanogrel 120 mg Then Placebo Then Temanogrel 60mg | Temanogrel 60 mg Then Temanogrel 120 mg Then Placebo | Temanogrel 60 mg Then Placebo Then Temanogrel 120 mg | Placebo Then Temanogrel 120 mg Then Temanogrel 60 mg | Placebo Then Temanogrel 60 mg Then Temanogrel 120 mg
Started | 2 | 2 | 2 | 2 | 3 | 2
Completed | 2 | 2 | 2 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants, irrespective of whether they received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Temanogrel 120 mg Then Temanogrel 60 mg Then Placebo | Temanogrel 120 mg Then Placebo Then Temanogrel 60mg | Temanogrel 60 mg Then Temanogrel 120 mg Then Placebo | Temanogrel 60 mg Then Placebo Then Temanogrel 120 mg | Placebo Then Temanogrel 120 mg Then Temanogrel 60 mg | Placebo Then Temanogrel 60 mg Then Temanogrel 120 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3 | 2 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 2 | 3 | 2 | 11
  >=65 years | 1 | 0 | 1 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 3 | 1 | 11
  Male | 0 | 1 | 0 | 0 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 2 | 3 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 2
  White | 2 | 2 | 1 | 2 | 2 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Digital Blood Flow Based on Rewarming Area Under the Curve (AUC) During Thirty Minutes Following a Cold Challenge
Description: Area under the curve for rewarming of digital blood flow after 30 minutes following a cold challenge was assessed. Area under the curve was defined as the area under the skin temperature curve and rewarming was a delicate phase of therapeutic hypothermia (TH). A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments for 30 minutes. Rewarming was assessed by infrared (IR) thermography which was an indirect method for evaluation of blood flow based on imaging skin temperature. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: FAS included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Degrees celsius*seconds
Groups:
- Temanogrel 120 mg: Participants received temanogrel 120 mg in the study.
- Temanogrel 60 mg: Participants received temanogrel 60 mg in this study.
- Placebo: Participants received placebo in this study.
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Degrees celsius*seconds | 43912 (4399.5) | 44000 (5308.2) | 44530 (8109.4)

2. Primary Outcome: Change in Digital Blood Flow Based on Reperfusion AUC During the Thirty Minutes Following a Cold Challenge
Description: Area under the curve for reperfusion of digital blood flow after 30 minutes following a cold challenge was assessed. A cold challenge was conducted by immersing hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments for 30 minutes. Reperfusion was assessed with laser speckle contrast imaging (LSCI) which was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. LSCI therefore provides quantitative measures of blood flow within predefined region of interests (ROIs) as mean arbitrary perfusion units, pu. Higher values of pu (and also pu*seconds) are considered better in the context of this trial. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: FAS included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Perfusion units*seconds
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Perfusion units*seconds | 118521 (99257.5) | 120748 (106766.5) | 147558 (144265.3)

3. Secondary Outcome: Maximum Reduction in Temperature Following a Cold Challenge Assessed With Infrared (IR) Thermography
Description: IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature. A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments for 30 minutes. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: FAS included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Degree Celsius | 23.06 (1.455) | 22.77 (1.770) | 22.45 (2.561)

4. Secondary Outcome: Maximum Reduction in Perfusion Temperature Following a Cold Challenge With Laser Speckle Contrast Imaging (LSCI)
Description: A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments for 30 minutes. LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. LSCI therefore provides quantitative measures of blood flow within predefined region of interests (ROIs) as mean arbitrary perfusion units, pu. Higher values of pu are considered better in the context of this trial. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: FAS included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Perfusion units | 33.67 (31.574) | 30.77 (30.898) | 36.04 (39.275)

5. Secondary Outcome: Maximum Recovery in Temperature Following a Cold Challenge Assessed With IR Thermography
Description: IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature. Changes in skin temperature at each visit were imaged IR thermography. A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments for 30 minutes. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: FAS included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Degree Celsius | 25.11 (2.863) | 25.38 (3.541) | 25.76 (5.080)

6. Secondary Outcome: Maximum Recovery in Perfusion Temperature Following a Cold Challenge Assessed With LSCI
Description: A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments for 30 minutes. LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. Changes in skin temperature at each visit were imaged using LSCI. LSCI therefore provides quantitative measures of blood flow within predefined region of interests (ROIs) as mean arbitrary perfusion units, pu. Higher values of pu are considered better in the context of this trial. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: FAS included all randomized participants, irrespective of whether they received any study treatment.
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Perfusion units | 137.9 (65.00) | 141.9 (70.47) | 159.6 (108.87)

7. Secondary Outcome: AUC During the Initial Two Minutes Following a Cold Challenge Assessed With IR Thermography
Description: AUC was defined as the area under the skin temperature curve. IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature. A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: Initial 2 minutes following a cold challenge
Population: FAS included all randomized participants, irrespective of whether they received any study treatment. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Degree Celsius*seconds
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Degree Celsius*seconds | 2830 (193.5) | 2792 (231.6) | 2741 (327.6)

8. Secondary Outcome: Perfusion AUC During the Initial Two Minutes Following a Cold Challenge Assessed With LSCI
Description: A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments. LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. LSCI therefore provides quantitative measures of blood flow within predefined region of interests (ROIs) as mean arbitrary perfusion units, pu. Higher values of pu (and also pu*seconds) are considered better in the context of this trial. AUC was defined as the area under the skin temperature curve, based on the LSCI results. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: Initial 2 minutes following a cold challenge
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Perfusion units*seconds
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Perfusion units*seconds | 7353 (4349.9) | 6959 (5093.5) | 6384 (5473.9)

9. Secondary Outcome: Slope During the Initial 2 Minutes (120 Seconds) Following a Cold Challenge Assessed With IR Thermography
Description: IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature. A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for 60 seconds, followed by post-cold challenge digital blood flow assessments. Slope was calculated based on the changes in skin temperature imaged using LSCI and IR thermography during the initial 120 seconds following the cold challenge. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: Initial 2 minutes following a cold challenge
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degree Celsius/seconds
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Degree Celsius/seconds | 0.203 (0.1786) | 0.212 (0.2900) | 0.251 (0.2922)

10. Secondary Outcome: Perfusion Slope During the Initial 2 Minutes (120 Seconds) Following a Cold Challenge Assessed With LSCI
Description: A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for 60 seconds, followed by post-cold challenge digital blood flow assessments. LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. LSCI therefore provides quantitative measures of blood flow within predefined region of interests (ROIs) as mean arbitrary perfusion units, pu. Higher values of pu (and also pu/seconds) are considered better in the context of this trial. Slope was calculated based on the changes in skin temperature imaged using LSCI during the initial 120 seconds following the cold challenge. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: Initial 2 minutes following a cold challenge
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Perfusion units/seconds
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Perfusion units/seconds | -6.437 (9.5172) | -0.841 (14.1211) | 0.652 (11.2937)

11. Secondary Outcome: Time to Achieve 50 Percent (%) Recovery From the Cold Challenge-Induced Reduction Assessed With IR Thermography and With LSCI
Description: IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature, while LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments. If 50% recovery was not achieved, the recovery time was set to 30 minutes. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Minutes
  IR thermography | 27.06 (6.78) | 25.70 (9.12) | 23.07 (10.72)
  LSCI: number analyzed (Participants) | 13 | 12 | 13
  LSCI | 10.68 (8.59) | 9.52 (6.61) | 3.98 (3.63)

12. Secondary Outcome: Time to Achieve 70 % Recovery From the Cold Challenge-Induced Reduction Assessed With IR Thermography and With LSCI
Description: IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature, while LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. A cold challenge was conducted by immersing the hands in a temperature-controlled water bath (15 [+/- 1] degree celsius) for one minute, followed by post-cold challenge digital blood flow assessments. If 70% recovery was not achieved, the recovery time was set to 30 minutes. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 30 minutes following a cold challenge
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Minutes
  IR thermography | 28.21 (5.01) | 26.24 (8.95) | 24.53 (10.18)
  LSCI: number analyzed (Participants) | 13 | 12 | 13
  LSCI | 12.99 (9.70) | 13.18 (7.27) | 5.34 (4.53)

13. Secondary Outcome: Change From Predose to Post-dose in Room Temperature Values as Assessed With IR Thermography
Description: IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature. Digital blood flow was assessed at each treatment visit at Predose for 5 minutes at room temperature, and at post-dose prior to cold challenge for 5 minutes at room temperature. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 5 minutes pre-dose, 5 minutes post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Degree Celsius | 0.576 (3.3539) | -0.278 (2.6927) | -0.803 (2.0125)

14. Secondary Outcome: Change From Predose to Post-dose in Room Temperature Perfusion Values as Assessed With LSCI
Description: Digital blood flow was assessed at each treatment visit at Predose for 5 minutes at room temperature, and at post-dose prior to cold challenge for 5 minutes at room temperature. LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. LSCI therefore provides quantitative measures of blood flow within predefined region of interests (ROIs) as mean arbitrary perfusion units, pu. Higher values of pu are considered better in the context of this trial. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 5 minutes pre-dose, 5 minutes post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Perfusion units | -0.01 (74.996) | -10.13 (68.037) | -50.16 (65.169)

15. Secondary Outcome: Change From Predose to Post-dose in Distal Dorsal Difference (DDD), Assessed With IR Thermography
Description: The distal dorsal difference was defined as the difference in temperature between the dorsum and the finger, from pre dose of study treatment to post-dose. IR thermography was an indirect method for evaluation of blood flow based on imaging skin temperature. Digital blood flow was assessed at each treatment visit at Predose for 5 minutes at room temperature, and at postdose prior to cold challenge for 5 minutes at room temperature. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 5 minutes pre-dose, 5 minutes post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Degree Celsius | -0.424 (1.7483) | -0.127 (1.7076) | 0.332 (1.5891)

16. Secondary Outcome: Change From Predose to Post-dose in Distal Dorsal Difference (DDD) [Perfusion], Assessed With LSCI
Description: Digital blood flow was assessed at each treatment visit at Predose for 5 minutes at room temperature, and at postdose prior to cold challenge for 5 minutes at room temperature. LSCI was based on differences in the speckle pattern (occurring when laser light illuminates a tissue) due to movement of blood cells. LSCI therefore provides quantitative measures of blood flow within predefined region of interests (ROIs) as mean arbitrary perfusion units, pu. Higher values of pu are considered better in the context of this trial. The distal dorsal difference was defined as the difference in perfusion temperature between the dorsum and the finger, from pre dose of study treatment to post-dose. Results presented were based on the average across all 8 fingers assessed (left index, left middle, left ring, left little, right index, right middle, right ring, right little).
Time Frame: 5 minutes pre-dose, 5 minutes post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Perfusion units
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Perfusion units | 3.56 (56.143) | 14.16 (57.611) | 34.86 (52.792)

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event was any untoward medical occurrence that did not necessarily have a causal relationship with study treatment. TEAE was an AE that occurred after initiation of study treatment that was not present at the time of treatment start or an AE that increased in severity after the initiation of medication, if the event was present at the time of treatment start. SAE was an AE resulting in any of the following outcomes or considered medically significant: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or birth defect.
Time Frame: Day 1 of dose to maximum of 4 (+/-1) days after last dose (up to maximum of 22 days)
Population: Safety set included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Temanogrel 60 mg: Participants received temanogrel 60 mg in the study.
- Placebo: Participants received placebo in the study.
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Participants
  TEAEs | 4 | 3 | 6
  Serious TEAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 of dose to maximum of 4 (+/-1) days after last dose (up to maximum of 22 days)
Arm/Group | Temanogrel 120 mg | Temanogrel 60 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 4/13 | 3/13 | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Temanogrel 120 mg (N=13) | Temanogrel 60 mg (N=13) | Placebo (N=13)
Headache (Nervous system disorders) | 1 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to a business decision that was not due to any safety concerns. The number of participants was smaller than originally planned and only summary statistics were therefore generated for primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT04915950/Prot_SAP_000.pdf